CLINICAL TRIAL: NCT06682923
Title: Evaluation of the MolecuLightDX Device in the Measurement of Surface Wounds in Patients
Brief Title: MolecuLightDX Measurement Feature Clinical Validation
Status: Recruiting | Type: Observational
Sponsor: MolecuLight Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 24-002
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-09

CONDITIONS: Wounds; Wound of Skin
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: MolecuLight DX Imaging Device — The MolecuLight DX Imaging Device is a fluorescence imaging device intended to acquire images from wounds. This will not alter the participant's standard of care treatment.

SUMMARY:
This is a prospective, single-arm, paired clinical evaluation of the MolecuLightDX device in the measurement of surface wounds in patients.

DETAILED DESCRIPTION:
The study compares the accuracy of wound measurements (area, length, and width) obtained using the ruler (standard of care) method and the MolecuLightDX device with a ground truth measurement (reference standard) derived from an expert panel.

ELIGIBILITY:
Inclusion Criteria:

* Willing to consent
* Willing to comply with all study procedures and availability for the duration of the study
* Male or female, aged over 22 years old
* Presented with diabetic foot ulcers, venous, arterial and pressure ulcers
* Wound size is greater than 0.5 cm2
* The wound has well-defined wound borders

Exclusion Criteria:

* Circumferential wound
* Wound without clearly defined wound borders
* Wound located in a difficult to reach/measure location
* Any contra-indication to routine wound care and/or monitoring
* Wounds with a length greater than 18.5cm or a width greater than 13.5cm.
* Tunneled or undermined wounds

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults 22 years and older with surface wounds
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Mean and SD of percent error for wound area by the MLI device in manual and automatic modes and by ruler | up to 6 months

SECONDARY OUTCOMES:
Mean and standard deviation of inter- and intra-user coefficient of variation (CV) for wound area measured by the MolecuLight device in manual and automaitc modes | up to 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - The Mayer Institute, Hamilton, Ontario
  - SHN Research Institute, Scarborough Village, Ontario

IPD SHARING:
Plan to Share IPD: Undecided